CLINICAL TRIAL: NCT03666156
Title: The Influence of Nutrition, Childhood and Adult Lifestyle Factors and Genetic Predisposition on Body Mass Index
Brief Title: Adult Weight, Genetics and Lifestyle Factors
Status: Completed | Type: Observational
Sponsor: St Mary's University College (Other)
Responsible Party: Sponsor
Other Study IDs: SMEC_2017-18_141
Record Dates: First submitted 2018-09-10; First posted 2018-09-11 (Actual); Last update posted 2018-12-07 (Actual); Status verified 2018-12

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Whole Sample: Female, caucasians, aged 18-65 years
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No Intervention

SUMMARY:
Childhood obesity leads to adulthood obesity, demonstrated in many retrospective and longitudinal studies. Genetics as a predictor of obesity is less established. Morandi et al, (2012) assessed whether lifestyle and genetic factors can be used to predict childhood obesity, concluding that genetics had minimal predictive effect. More recently Seyednasrollah, (2017) demonstrated that genetic information, when alongside clinical factors for cardiovascular disease, increased the predictive accuracy of obesity risk in adults. This study aims to investigate if known lifestyle and genetic risk factors are associated with BMI and if they can be used as predictors of overweight/obesity in adults.

ELIGIBILITY:
Inclusion Criteria:

* European Citizen.
* Aged between 18-65 years.
* Female.
* Caucasian

Exclusion Criteria:

* Currently following a diet or weight loss plan or have not been for over 6 months of the previous year.
* Suffering from diabetes (type I or II).
* Cancer, or have had cancer in the past.

Ages: 18 Years to 65 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: European Citizen Aged between 18-65 years Female. Caucasian
Sampling Method: Non-Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2018-12-06 (Actual); Study Completion 2018-12-06 (Actual)

PRIMARY OUTCOMES:
Body Mass Index | September - November 2018

CONTACTS AND LOCATIONS:
Locations (1):
- St Mary's University, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No